CLINICAL TRIAL: NCT07131033
Title: Effects of Perioperative Intravenous Infusion Esketamine Combined With Magnesium Sulfate for Postoperative Fatigue Syndrome in Patients Undergoing Laparoscopic Cholecystectomy: A 2×2 Factorial Randomized Controlled Trial
Brief Title: Esketamine Combined With Magnesium Sulfate for Postoperative Fatigue Syndrome in Patients Undergoing Laparoscopic Cholecystectomy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second People's Hospital of Huai'an (Other)
Responsible Party: Principal Investigator, Chenglan Xie, chief physician, The Second People's Hospital of Huai'an
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLanXie
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Cholecystectomy; Alleviate Postoperative Fatigue Syndrome
Keywords: esketamine; magnesium sulfate; postoperative fatigue syndrome; Laparoscopic Cholecystectomy
MeSH Terms: interventions — Esketamine; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization sequence was generated by a computer and handed over in sealed opaque sequentially numbered envelopes. The envelope was opened by anaesthetist not involved in the study and drugs were dispensed as per the allocation card. The configured drugs were then handed over to experienced anaesthetists who were not aware of the subgroups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Esketamine (Experimental): Patients were given intravenous esketamine 0.25 mg/kg 10 min before induction of anaesthesia, followed by continuous pumping at 0.25 mg/(kg-h) until the end of the operation.
  Interventions: Drug: Esketamine
- Magnesium Sulfate (Experimental): Patients were injected with 30 mg/kg of magnesium sulphate intravenously 10 min before the induction of anaesthesia, followed by continuous pumping at 10 mg/(kg-h) until the end of the operation.
  Interventions: Drug: Magnesium sulfate
- Esketamine and Magnesium Sulfate (Experimental): Patients received a simultaneous intravenous infusion of esketamine (0.25 mg/kg) and magnesium sulfate (30 mg/kg) over 10 minutes before anesthesia induction, followed by continuous infusion of esketamine at 0.25 mg/kg/h and magnesium sulfate at 10 mg/kg/h via separate channels until surgery completion.
  Interventions: Drug: Esketamine and Magnesium sulfate
- Control (Placebo Comparator): Patients in the control group received an equivalent volume of normal saline infused intravenously over 10 minutes before anesthesia induction, followed by continuous saline infusion at a matched flow rate via a separate channel until surgery completion.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esketamine — Patients were given intravenous esketamine 0.25 mg/kg 10 min before induction of anaesthesia, followed by continuous pumping at 0.25 mg/(kg-h) until the end of the operation.
  Arms: Esketamine
Drug: Magnesium sulfate — Patients were injected with 30 mg/kg of magnesium sulphate intravenously 10 min before the induction of anaesthesia, followed by continuous pumping at 10 mg/(kg-h) until the end of the operation.
  Arms: Magnesium Sulfate
Drug: Esketamine and Magnesium sulfate — Patients received a simultaneous intravenous infusion of esketamine (0.25 mg/kg) and magnesium sulfate (30 mg/kg) over 10 minutes before anesthesia induction, followed by continuous infusion of esketamine at 0.25 mg/kg/h and magnesium sulfate at 10 mg/kg/h via separate channels until surgery completion.
  Arms: Esketamine and Magnesium Sulfate
Drug: Saline — Patients in the control group received an equivalent volume of normal saline infused intravenously over 10 minutes before anesthesia induction, followed by continuous saline infusion at a matched flow rate via a separate channel until surgery completion.
  Arms: Control

SUMMARY:
Laparoscopic cholecystectomy (LC), while minimally invasive, triggers postoperative fatigue syndrome (POFS) through mechanisms including ischemia-reperfusion injury, neuroendocrine stress (sustained cortisol elevation), and inflammation-driven mitochondrial dysfunction (IDO-mediated kynurenine production). Esketamine, an NMDA receptor antagonist, counteracts POFS by blocking central sensitization, suppressing neuroinflammation (e.g., microglial IL-6 release), and enhancing neuroplasticity via BDNF/TrkB upregulation. Magnesium sulfate complements this by antagonizing NMDA/voltage-gated calcium channels to reduce inflammation and calcium overload, while optimizing cellular energy metabolism as an ATPase cofactor and alleviating muscle spasms. Crucially, their combination holds synergistic potential: esketamine targets central fatigue pathways, while magnesium addresses peripheral metabolic and muscular components. This study aims to determine their individual and interactive effects on POFS, recovery quality, and sleep outcomes in LC patients, establishing an efficient, safe strategy to accelerate postoperative rehabilitation.

DETAILED DESCRIPTION:
This randomized, double-blind trial investigated the effects of esketamine and magnesium sulfate on postoperative fatigue syndrome in patients undergoing laparoscopic cholecystectomy. Using computer-generated randomization and sealed envelopes, 120 patients were allocated in a 1:1:1:1 ratio to four groups: Group E received intravenous esketamine (0.25 mg/kg over 10 min pre-induction followed by 0.25 mg/kg/h); Group M received magnesium sulfate (30 mg/kg over 10 min pre-induction followed by 10 mg/kg/h); Group EM received both drugs concurrently at the specified doses; and Group C received volume-matched normal saline. Patients, attending anesthesiologists, and outcome assessors remained blinded to group assignment throughout the study, with intraoperative management handled by a separate non-investigating anesthesiologist to preserve blinding integrity.

The patients were routinely fasted for 6 h and abstained from drinking for 2 h preoperatively. All patients were not anesthetized with premedication. After admission, patients were routinely administered oxygen by mask, peripheral venous access was opened and cardiac monitoring, including noninvasive blood pressure, pulse oximetry, electrocardiogram, body temperature and entropy index, was routinely performed. Both groups were routinely rapidly induced with midazolam 0.05 mg/kg, propofol 1.5 mg/kg, rocuronium bromide 1mg/kg, and sufentanil 0.5 μg/kgrespectively. Preoxygenation was administered for 3 min followed by endotracheal intubation and connection to a ventilator with 50％ oxygen of 2.0 L/min for respiratory control. Setting parameters: tidal volume 6～8 ml/kg, inspiratory ratio 1:2, control PETCO2 at 35～40 mmHg. During anaesthesia maintenance, remifentanil 0.1-0.5 ug/kg/min, sevoflurane (1%-3%) and propofol 4-12 mg/kg/h were continuously infused in all three groups.Sevoflurane (1%-3%), and Propofol 4-12 mg/kg/h were continuously infused in all three groups.A four-channel microinfusion pump was used for synchronous intravenous infusion. Each drug was administered through an independent channel to avoid drug interactions, and the drugs were continuously infused during the operation until the end of the surgery. The appropriate depth of anesthesia (entropy index RE/SE 40-60) was maintained by adjusting the infusion rate of propofol and remifentanil. At the appropriate depth of anaesthesia, vasoactive drugs (ephedrine, phenylephrine, nitroglycerin) can be administered to regulate blood pressure.After the operation, the patient was immediately transferred to the PACU. when the patient regained consciousness and could breathe on his own, the tracheal tube was removed. In the PACU, 30 mg of ketorolac tromethamine was administered intravenously to relieve analgesia if the patient's NRS score was >3 or if the patient required analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) classification I-II
* Patients scheduled for LC under general anaesthesia and with a procedure duration of less than 60 minutes.

Exclusion Criteria:

* Patients who do not sign the informed consent;
* patients with severe diseases of major organs such as the heart, brain, lungs, liver, and kidneys;
* patients with adverse drug reactions to esketamine or magnesium sulfate;
* patients with uncontrolled hypertension or hyperthyroidism;
* patients with endocrine and metabolic diseases or neurological diseases;
* pregnant or lactating women;
* long-term users of sedatives, analgesics, or long-term alcohol abusers;
* patients with a history of mental illness, language communication barriers, or inability to understand the content of the experiment;
* patients with difficult airways during anesthesia induction requiring a change in the conventional intubation method;
* patients with sinus bradycardia or atrioventricular block;
* patients with concurrent cholangitis, biliary obstruction, or pancreatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Christensen's Fatigue Scale | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 2 (POD2), postoperative day 7 (POD7), postoperative day 30 (POD30)
  The Christensen Fatigue Scale, a widely used unidimensional tool for assessing postoperative fatigue syndrome, relies on patients' subjective ratings of fatigue and daily activity ability on a 1-10 scale, with no multiple subdimensions or specific items. Scoring criteria are: 1-2 points (normal, fatigue only with excessive activity, normal sleep); 3-5 points (able to perform daily activities, occasional slightly strenuous activity); 6-8 points (maintaining only partial daily activities, difficulty with walking/climbing stairs, need for sleep); 9-10 points (unable to perform daily activities, extreme need for sleep). A score > 2 points indicates fatigue, while ≥ 6 points may signal clinically noticeable postoperative fatigue syndrome.
Identity-Consequence Fatigue Scale | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 2 (POD2), postoperative day 7 (POD7), postoperative day 30 (POD30)
  The 31-item Identity-Consequence Fatigue Scale (ICFS), which is a multidimensional self-report questionnaire designed to comprehensively assess fatigue, captures fatigue's complexity by exploring its interactions with one's sense of identity and consequent impacts on daily functioning, emotional states, and social interactions. For scoring, items typically use Likert-type scales (with slight variations in response options across items), some requiring reverse scoring for consistent interpretation. Total scores are summed, with the minimum and maximum values of the total score to be specified based on the scale's scoring criteria; higher scores indicate more severe (worse) fatigue. This comprehensive 31-item structure enables detailed exploration of fatigue, suiting research needing a thorough understanding of its multifaceted nature.

SECONDARY OUTCOMES:
The Quality of Recovery-15（QoR-15） | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 2 (POD2)
  The QoR-15 scale is divided into five dimensions: physical comfort (5 items), self-care (2 items), psychological support (2 items), emotional state (4 items), and pain (2 items), with each item rated on a scale of 0-10, and the total score ranging from 0-150, with the higher the score the better the quality of recovery, and a score of 118 and above indicating surgery.
Numeric Rating Scale（NRS） | 5 minutes after extubation, postoperative day 1 (POD1), postoperative day 2 (POD2)
  NRS is a rating used to assess a patient's level of pain, which is assessed by the patient based on self-perception on a scale from 0 to 10. A score of 0 represents no pain and a score of 10 represents the most pain.
Richmond Agitation and Sedation Scale(RASS) | 5 minutes after extubation, postoperative day 1 (POD1), postoperative day 2 (POD2)
  The Richmond Agitation-Sedation Scale (RASS) is a widely used tool to assess the level of sedation and agitation in patients. It ranges from +4 to -5, with specific descriptors for each score: +4 indicates combative behavior; +3 is extremely agitated; +2 means agitated and restless ; +1 denotes restless but calm; 0 represents alert and calm; -1 is drowsy; -2 indicates light sedation; -3 means moderate sedation; -4 is deep sedation ; and -5 represents unarousable. This scale helps clinicians objectively evaluate and adjust sedation levels to ensure patient comfort and safety.
Mean arterial blood pressure(MAP) | Perioperative:entering the operating room, before induction of anesthesia, before intubation, immediately after intubation, start of surgery, end of surgery, at extubation
  perioperative hemodynamic fluctuations
sleep duration | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 2 (POD2)
  Sleep data such as sleep duration recorded by actigraphs.
grip strength | Preoperative day 1 (PRE1), postoperative day 1 (POD1), postoperative day 2 (POD2)
  The electronic dynamometer measures grip strength.
Discontinuation time, extubation time | Postoperative
  Patient awakening time and extubation time (time from stopping medication to awakening and extubation)
Drug use | Perioperative
  The names and dosages of the patients' intraoperative anaesthetic drugs (propofol and remifentanil), vasoactive drugs, and postoperative analgesic drugs were recorded.
Incidence of adverse reactions | postoperative day 1 (POD1), postoperative day 2 (POD2)
  respiratory depression, postoperative coughing, incidence of postoperative nausea and vomiting, postoperative hoarseness, sore throat, hallucinations, drowsiness, nightmares, blurred vision, sensory abnormalities, dissociative symptoms, cognitive decline, muscle strength reduction

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Huaian Hospital of Xuzhou Medical University, Huai'an Second Hospital, Huaian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacourt TE, Vichaya EG, Chiu GS, Dantzer R, Heijnen CJ. The High Costs of Low-Grade Inflammation: Persistent Fatigue as a Consequence of Reduced Cellular-Energy Availability and Non-adaptive Energy Expenditure. Front Behav Neurosci. 2018 Apr 26;12:78. doi: 10.3389/fnbeh.2018.00078. eCollection 2018. PMID 29755330
- [Background] Zargar-Shoshtari K, Hill AG. Postoperative fatigue: a review. World J Surg. 2009 Apr;33(4):738-45. doi: 10.1007/s00268-008-9906-0. PMID 19189174
- [Background] Zhuang CL, Mao XY, Liu S, Chen WZ, Huang DD, Zhang CJ, Chen BC, Shen X, Yu Z. Ginsenoside Rb1 improves postoperative fatigue syndrome by reducing skeletal muscle oxidative stress through activation of the PI3K/Akt/Nrf2 pathway in aged rats. Eur J Pharmacol. 2014 Oct 5;740:480-7. doi: 10.1016/j.ejphar.2014.06.040. Epub 2014 Jun 27. PMID 24975098
- [Background] Chen W, Liu S, Chen F, Zhou C, Zhuang C, Shao S, Yu J, Huang D, Chen B, Yu Z. [Relationship between NMDA receptor and postoperative fatigue syndrome and its associated central mechanism]. Zhonghua Wei Chang Wai Ke Za Zhi. 2015 Apr;18(4):376-81. Chinese. PMID 25940183
- [Background] Wang X, Lin C, Lan L, Liu J. Perioperative intravenous S-ketamine for acute postoperative pain in adults: A systematic review and meta-analysis. J Clin Anesth. 2021 Feb;68:110071. doi: 10.1016/j.jclinane.2020.110071. Epub 2020 Oct 26. PMID 33007645
- [Background] Lin X, Feng X, Sun L, Wang Y, Wu X, Lu S, Shao L, Wang W, Yang L, Geng W, Lin H. Effects of esketamine on postoperative fatigue syndrome in patients after laparoscopic resection of gastric carcinoma: a randomized controlled trial. BMC Anesthesiol. 2024 May 24;24(1):185. doi: 10.1186/s12871-024-02513-w. PMID 38789968
- [Background] Sun L, Zhao Y, Li Y, Zhai W, Gao F, Yin Q, Cheng W, Wang Z, Zeng Y. Effect of continuous subanesthetic esketamine infusion on postoperative fatigue in patients undergoing laparoscopic radical resection for colorectal cancer: a randomized controlled study. Am J Cancer Res. 2023 Jun 15;13(6):2554-2563. eCollection 2023. PMID 37424809
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Fritzen R, Davies A, Veenhuizen M, Campbell M, Pitt SJ, Ajjan RA, Stewart AJ. Magnesium Deficiency and Cardiometabolic Disease. Nutrients. 2023 May 17;15(10):2355. doi: 10.3390/nu15102355. PMID 37242238